CLINICAL TRIAL: NCT00191152
Title: Randomized Trial of Gemcitabine Plus Docetaxel vs. Docetaxel Plus Capecitabine in Metastatic Breast Cancer in 1st and 2nd
Brief Title: A Phase III Trial For Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4703; B9E-US-S188
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-12-08 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer; Breast Neoplasms; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine + Docetaxel (Experimental)
  Interventions: Drug: gemcitabine; Drug: docetaxel
- Capecitabine + Docetaxel (Active Comparator)
  Interventions: Drug: docetaxel; Drug: capecitabine

INTERVENTIONS:
Drug: gemcitabine — 1000 mg/m2, intravenous (IV) day 1 and day 8 every 21 days until disease progression
  Other Names: LY188011; Gemzar
  Arms: Gemcitabine + Docetaxel
Drug: docetaxel — 75 mg/m2, intravenous (IV), every 21 days until disease progression
Drug: capecitabine — 1000 mg/m2, by mouth (PO) twice a day (BID), days 1-14, every 21 days until disease progression
  Arms: Capecitabine + Docetaxel

SUMMARY:
This is a phase III randomized study between the docetaxel/gemcitabine and docetaxel/ capecitabine doublets, with crossover to the alternate agent. The experimental arm will receive gemcitabine 1000 mg/m2 intravenous (IV) over 30 minutes days 1 and 8 and docetaxel 75 mg/m2 IV day 1 over 1 hour repeated every three weeks. The comparator arm will receive docetaxel 75 mgm/m2 IV day 1 over 1 hour and oral capecitabine 1000 mg/m2 twice daily, days 1 through 14 repeated every three weeks. Patients who progress on the experimental arm, will be treated with capecitabine as dosed on the comparator arm. Patients who progress on the comparator arm will be treated with gemcitabine as dosed on the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of breast cancer with locally advanced and/or metastatic disease
* Patients may have received prior neo-adjuvant or adjuvant taxane regimen as long as it has been greater than or equal to 6 months since completion of the regimen
* Patients may have had 0-1, but no more than one prior course of chemotherapy for metastatic disease
* Patients must have either measurable or non-measurable (evaluable) disease
* Prior radiation therapy allowed of less than 25% of the bone marrow

Exclusion Criteria:

* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated at least 5 years previously with no evidence of recurrence)
* Parenchymal or leptomeningeal brain metastases
* Peripheral neuropathy greater than or equal to grade 2
* Prior treatment with gemcitabine and capecitabine will not be allowed. Prior treatment with a taxane in the metastatic setting will not be allowed. Prior taxane therapy in the neo-adjuvant or adjuvant setting is allowed if completion of therapy greater than or equal to 6 months prior to enrollment.
* Active cardiac disease not controlled by therapy and/or myocardial infarction within the preceding 6 months.
* Concomitant Herceptin is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2002-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (65):
- United States (47):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Fort Smith, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Hot Springs, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Springdale, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Berkeley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Fountain Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Highland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Rancho Mirage, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Santa Rosa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Sylmar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Torrington, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Royal Oak, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Southfield, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Fremont, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Voorhees Township, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Springfield, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician.c, Dunmore, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Franklin, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Johnstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Kittanning, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Madison, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Capital Federal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Mendoza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Santa Fe
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Waratah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Redcliffe, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Ashford, South Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Porto Alegre, Brazil
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Acapulco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Michoacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Toluca
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Taoyuan District

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not all participants who completed initial treatment went on to crossover treatment. Per protocol, participants had the option to go off study without receiving crossover treatment.
Groups:
- Gemcitabine Plus Docetaxel: Initial treatment: Gemcitabine 1000 milligrams per meter squared (mg/m2),intravenous (IV) on Days 1 and 8 every 21 days plus docetaxel 75 mg/m2 IV on Day 1 every 21 days. This treatment continues until progression of disease (PD), at which time crossover treatment begins.
  Crossover treatment: capecitabine 1000 mg/m2 by mouth (PO) twice a day (BID), Days 1-14, every 21 days until PD at which time all treatment is discontinued. PD during crossover was defined as the Response Evaluation Criteria in Solid Tumors (RECIST) guideline with the tumor measurement at the start of crossover treatment (or end of initial treatment) considered as the crossover baseline, with subsequent tumor measurements during crossover treatment compared to the crossover baseline.
- Docetaxel Plus Capecitabine: Initial treatment: Docetaxel 75 milligrams per meter squared (mg/m2), intravenous (IV) on Day 1 every 21 days plus capecitabine 1000 mg/m2, by mouth (PO), twice a day (BID), Days 1-14, every 21 days. This treatment continues until progression of disease (PD), at which time crossover treatment begins.
  Crossover treatment: gemcitabine 1000 mg/m2, IV, Days 1 and 8, every 21 days. This treatment continues until PD at which time all treatment is discontinued.
Period: Initial Treatment
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Started | 239 | 236
Received Initial Treatment | 236 | 227
Completed | 98 | 83
Not Completed | 141 | 153
Not completed — Adverse Event | 43 | 67
Not completed — Physician Decision | 40 | 31
Not completed — Withdrawal by Subject | 40 | 28
Not completed — Lost to Follow-up | 0 | 6
Not completed — Other | 18 | 21
Period: Crossover Treatment
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Started | 77 | 81
Received Treatment | 76 | 80
Completed | 50 | 53
Not Completed | 27 | 28
Not completed — Adverse Event | 8 | 8
Not completed — Physician Decision | 7 | 7
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine Plus Docetaxel: Initial treatment: Gemcitabine 1000 milligrams per meter squared (mg/m2), intravenous (IV) on Days 1 and 8 every 21 days plus docetaxel 75 mg/m2 IV on Day 1 every 21 days. This treatment continues until progression of disease (PD), at which time crossover treatment begins.
  Crossover treatment: capecitabine 1000 mg/m2 by mouth (PO)twice a day (BID), Days 1-14, every 21 days until progressive disease (PD) at which time all treatment is discontinued.
- Docetaxel Plus Capecitabine: Initial treatment: Docetaxel 75 milligrams per meter squared (mg/m2), intravenous (IV) on Day 1 every 21 days plus capecitabine 1000 mg/m2, by mouth (PO), twice a day (BID),Days 1-14, every 21 days. This treatment continues until progression of disease (PD), at which time crossover treatment begins.
  Crossover treatment: gemcitabine 1000 mg/m2, IV, Days 1 and 8, every 21 days. This treatment continues until PD at which time all treatment is discontinued.
- Total: Total of all reporting groups
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine | Total
Number analyzed (Participants) | 239 | 236 | 475
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.77) | 54.6 (11.60) | 55.2 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 1 | 238
  Male | 2 | 235 | 237
Region of Enrollment [Number; unit: participants]
  United States | 173 | 166 | 339
  Taiwan | 15 | 18 | 33
  Mexico | 14 | 15 | 29
  Puerto Rico | 4 | 1 | 5
  Argentina | 11 | 13 | 24
  Brazil | 1 | 1 | 2
  Australia | 11 | 12 | 23
  Korea, Republic of | 10 | 10 | 20
Karnofsky Performance Status-Baseline [Number; unit: units on a scale] — Classifies patients according to their functional impairment. Scores range from 0-100, the lower the score, the worse the survival for most serious illnesses.
  units on a scale
    <=60 Needs increasing assistance up to Death (0) | 0 | 0 | 0
    70 - Unable to carry on normal activity | 16 | 15 | 31
    80 - Activity with effort; some signs of disease | 44 | 40 | 84
    90 - Normal activity; minor signs of disease | 101 | 101 | 202
    100 - Normal no complaints; no evidence of disease | 74 | 75 | 149
    Missing | 4 | 5 | 9
Race/Ethnicity [Number; unit: participants]
  Caucasian | 160 | 158 | 318
  African Descent | 23 | 12 | 35
  Oriental | 28 | 30 | 58
  Hispanic | 26 | 36 | 62
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Time to Disease Progression (Crossover Treatment)
Description: For crossover treatment, time to disease progression (TTDP) was defined as the number of months between the first dose date of crossover treatment and the date of disease progression or the date of death due to disease under study, whichever came first. TTDP for crossover treatment only applied to those participants who crossed over from initial treatment to crossover treatment. TTDP censored at earliest of: 1)date of death not due to disease; or 2)date of last contact for participants alive without disease progression; or 3)start date of other anti-tumor therapy due to progression.
Time Frame: Date of first dose of crossover treatment to date of first-documented disease progression after receiving first crossover treatment or date of death due to study disease, whichever came first (up to 82 months)
Population: ITT population: all randomized participants. Censored participants in crossover treatment: 13 in capecitabine arm; 10 in gemcitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Capecitabine: capecitabine 1000 mg/m2, by mouth two times per day, days 1-14 every 21 days until progression of disease at which time all treatment is discontinued.
- Gemcitabine: gemcitabine 1000 mg/m2, intravenous, days 1 and 8 every 21 days until progression of disease at which time all treatment is discontinued.
Arm/Group | Capecitabine | Gemcitabine
Number analyzed (Participants) | 77 | 81
months | 4.51 [2.11 to 7.80] | 2.34 [2.04 to 3.78]
Statistical Analysis 1: Comparison: Capecitabine vs Gemcitabine; Test type: Superiority or Other; p = 0.145, Log Rank

2. Secondary Outcome: Progression-Free Survival (Initial Treatment)
Description: For initial treatment, progression-free survival (PFS) was defined as the number of months between the date of randomization and the date of first documented disease progression or the date of death due to any cause, whichever came first. Time to PFS was censored at the earliest of: 1) date of last contact for participants alive without disease progression; or 2) start date of other anti-tumor therapy for progression; or 3) first dose date of crossover treatment.
Time Frame: Date of randomization until the date of first documented progression or date of death from any cause, whichever came first (up to 82 months)
Population: ITT: all randomized participants. Censored participants (initial treatment): 64 in gemcitabine/docetaxel arm; 80 in docetaxel/capecitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gemcitabine Plus Docetaxel: gemcitabine 1000 mg/m2, intravenous on days 1 and 8 every 21 days plus docetaxel 75 mg/m2 intravenous on day 1 every 21 days. This treatment continues until progression of disease at which time crossover treatment begins.
- Docetaxel Plus Capecitabine: docetaxel 75 mg/m2, intravenous, on day 1 every 21 days plus capecitabine 1000 mg/m2, by mouth twice a day, days 1-14, every 21 days. This treatment continues until progression of disease at which time crossover treatment begins.
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Number analyzed (Participants) | 239 | 236
months | 9.01 [7.73 to 10.53] | 8.88 [7.27 to 10.89]
Statistical Analysis 1: Comparison: Gemcitabine Plus Docetaxel vs Docetaxel Plus Capecitabine; Test type: Superiority or Other; p = 0.361, Log Rank

3. Secondary Outcome: Progression-Free Survival (Crossover Treatment)
Description: For crossover treatment, progression-free survival (PFS) was defined as the number of months between first dose date of crossover treatment and date of documented disease progression or date of death due to any cause, whichever came first. PFS for crossover treatment only applied to those participants who crossed over from initial treatment to crossover treatment. PFS was censored at the earliest of: 1) date of last contact for participants alive without disease progression; or 2) start date of other anti-tumor therapy for participants with documented disease progression.
Time Frame: First dose date of crossover treatment to date of first-documented progression after receiving crossover treatment or date of death due to any cause, whichever came first (up to 82 months)
Population: ITT population: all randomized participants. Censored participants, crossover treatment: 13 in capecitabine arm; 10 in gemcitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine | Gemcitabine
Number analyzed (Participants) | 77 | 81
months | 4.51 [2.11 to 7.80] | 2.34 [2.04 to 3.78]
Statistical Analysis 1: Comparison: Capecitabine vs Gemcitabine; Test type: Superiority or Other; p = 0.145, Log Rank

4. Primary Outcome: Time to Disease Progression (Initial Treatment)
Description: Time to disease progression (TTDP) at initial treatment was defined as the number of months between date of randomization and the date of first documented disease progression or the date of death due to disease under study, whichever came first. TTDP censored at earliest of: 1) date of death not due to disease; or 2) date of last contact for participants alive without disease progression; or 3) start date of other anti-tumor therapy; or 4) first dose date of crossover treatment.
Time Frame: Randomization date to the earliest date of first documented disease progression date or the date of death if the participant died due to study disease (up to 82 months)
Population: Intent-to-treat (ITT) population: all randomized participants. Censored participants in initial treatment: 68 gemcitabine/docetaxel arm; 83 docetaxel/capecitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gemcitabine Plus Docetaxel: gemcitabine 1000 milligrams per meter squared (mg/m2) intravenous, days 1 and 8 every 21 days plus docetaxel 75 mg/m2, intravenous, day 1 every 21 days.
  Treatment continues until progression of disease at which time crossover treatment begins.
- Docetaxel Plus Capecitabine: docetaxel 75 mg/m2, intravenous, day 1 every 21 days plus capecitabine 1000 mg/m2, by mouth twice a day, days 1-14 every 21 days. Treatment continues until progression of disease, at which time crossover treatment begins.
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Number analyzed (Participants) | 239 | 236
months | 9.28 [7.73 to 10.79] | 8.88 [7.37 to 11.05]
Statistical Analysis 1: Comparison: Gemcitabine Plus Docetaxel vs Docetaxel Plus Capecitabine; Test type: Superiority or Other; p = 0.385, Log Rank

5. Secondary Outcome: Duration of Response (Initial Treatment)
Description: Among tumor responders, duration of tumor response was measured from the date of response (complete response [CR] or partial response [PR] until the first date of documented progression or death from any cause. Duration of response was censored at the earliest of: 1) date of last contact for participants alive without disease progression (DP); or 2) start date of other anti-tumor therapy for DP; or 3) dose date of crossover treatment.
Time Frame: Date of response (CR or PR) until the first date of documented progression or death from any cause (up to 82 months)
Population: ITT population: participants with CR or PR as best overall response (initial treatment). Censored participants: 16 in gemcitabine/docetaxel arm; 30 in docetaxel/capecitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Number analyzed (Participants) | 77 | 85
months | 9.11 [7.60 to 11.94] | 10.39 [8.22 to 13.75]
Statistical Analysis 1: Comparison: Gemcitabine Plus Docetaxel vs Docetaxel Plus Capecitabine; Test type: Superiority or Other; p = 0.377, Log Rank

6. Secondary Outcome: Duration of Response (Crossover Treatment)
Description: At crossover treatment, duration of response was measured from the time criteria were met for complete response (CR) or partial response (PR), until first date that recurrent or progressive disease was objectively documented or date of death due to any cause, whichever came first. This definition only applied to those who crossed over & achieved CR or PR in crossover treatment. Duration of response censored at earliest of: 1) date of last contact for those alive without disease progression; or 2) start date of other anti-tumor therapy for documented disease progression.
Time Frame: Date of CR or PR until first date of recurrent or progressive disease after receiving crossover treatment was objectively documented or date of date due to any cause, whichever came first (up to 82 months)
Population: ITT population: participants with CR or PR as best overall response at crossover treatment. Censored participants: 4 in capecitabine arm; 2 in gemcitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine | Gemcitabine
Number analyzed (Participants) | 11 | 7
months | 25.89 [4.64 to 45.03] | 42.50 [16.02 to 48.22]
Statistical Analysis 1: Comparison: Capecitabine vs Gemcitabine; Test type: Superiority or Other; p = 0.446, Log Rank

7. Secondary Outcome: Overall Survival
Description: Overall survival time was defined as the number of months between the date of randomization and the date of death due to any cause. The overall survival time was censored at the date of last contact for participants who were still alive.
Time Frame: Date of randomization to date of death from any cause (up to 82 months)
Population: Intent to treat population: all randomized participant. Censored participants: 75 in gemcitabine/docetaxel arm; 72 in docetaxel/capecitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gemcitabine Plus Docetaxel: gemcitabine 1000 mg/m2, intravenous, days 1 and 8 every 21 days plus docetaxel 75 mg/m2, intravenous, day 1 every 21 days. Treatment continues until progression of disease at which time crossover treatment begins.
- Docetaxel Plus Capecitabine: docetaxel 75 mg/m2, intravenous, day 1 every 21 days plus capecitabine 1000 mg/m2, by mouth twice a day, days 1-14 every 21 days. Treatment continues until progression of disease at which time crossover treatment begins.
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Number analyzed (Participants) | 239 | 236
months | 22.99 [18.82 to 25.69] | 23.29 [18.55 to 25.53]
Statistical Analysis 1: Comparison: Gemcitabine Plus Docetaxel vs Docetaxel Plus Capecitabine; Test type: Superiority or Other; p = 0.785, Log Rank

8. Secondary Outcome: Best Overall Response (Initial Treatment)
Description: Best overall response was the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response was assessed using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that did not meet above criteria.
Time Frame: Best response from start of treatment until disease progression/recurrence (up to 82 months)
Population: ITT population.
Measure: Number; unit: participants
Groups:
- Docetaxel Plus Capecitabine: docetaxel 75 mg/m2, intravenous, day 1 every 21 days plus capecitabine 1000 mg/m2, by mouth twice a day, days 1-14, every 21 days. Treatment continues until progression of disease at which time crossover treatment begins.
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Number analyzed (Participants) | 239 | 236
participants
  Complete Response (confirmed) | 6 | 6
  Partial Response (confirmed) | 71 | 79
  Stable Disease | 96 | 90
  Progressive Disease | 32 | 27
  Unknown | 34 | 34
Statistical Analysis 1: Comparison: Gemcitabine Plus Docetaxel vs Docetaxel Plus Capecitabine; Test type: Superiority or Other; p = 0.364, Fisher Exact

9. Secondary Outcome: Best Overall Response (Crossover Treatment)
Description: Best overall response was the best response recorded from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response assessed using RECIST criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that did not meet above criteria.
Time Frame: Best response from start of treatment until disease progression/recurrence (up to 82 months)
Population: Only included participants who crossed over from initial treatment to crossover treatment.
Measure: Number; unit: participants
Arm/Group | Capecitabine | Gemcitabine
Number analyzed (Participants) | 77 | 81
participants
  Complete Response (confirmed) | 1 | 1
  Partial Response (confirmed) | 10 | 6
  Stable Disease | 19 | 20
  Progressive Disease | 34 | 36
  Unknown | 13 | 18
Statistical Analysis 1: Comparison: Capecitabine vs Gemcitabine; Test type: Superiority or Other; p = 0.446, Fisher Exact

10. Secondary Outcome: Summary of Changes in Karnofsky Performance Status (KPS) by Treatment (Initial Treatment)
Description: KPS ranges from 0 to 100, subdivided into three categories: incapacitated (0-40), self-care (50-70), and normal activity (80-100).
Time Frame: Baseline until crossover treatment began (up to 82 months)
Population: Intent-to-treat population, initial treatment, participants with KPS at baseline and end of initial treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Number analyzed (Participants) | 212 | 214
units on a scale
  Baseline | 90.85 (8.159) | 90.09 (8.335)
  Change from Baseline | -3.30 (9.259) | -3.27 (9.118)
Statistical Analysis 1: Comparison: Gemcitabine Plus Docetaxel vs Docetaxel Plus Capecitabine; Test type: Superiority or Other; p = 0.990, Mixed Models Analysis

11. Secondary Outcome: Summary of Changes in Karnofsky Performance Status (KPS) by Treatment (Crossover Treatment)
Description: as for outcome 10
Time Frame: First day of crossover treatment until end of crossover treatment at trial discontinuation (up to 82 moths)
Population: Participants with KPS at baseline (conclusion of initial treatment) and end of crossover treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Capecitabine: capecitabine 1000 mg/m2, by mouth two times per day, days 1-14, every 21 days
- Gemcitabine: gemcitabine 1000 mg/m2 intravenously, days 1 and 8, every 21 days
Arm/Group | Capecitabine | Gemcitabine
Number analyzed (Participants) | 66 | 63
units on a scale
  Baseline | 89.09 (7.174) | 87.94 (9.360)
  Change from Baseline | -0.30 (7.839) | -1.27 (9.068)
Statistical Analysis 1: Comparison: Capecitabine vs Gemcitabine; Test type: Superiority or Other; p = 0.117, Mixed Models Analysis

12. Secondary Outcome: Summary of Changes in Rotterdam Symptom Checklist (RSCL) by Treatment (Initial Treatment)
Description: RSCL includes 4 scales to assess quality of life (QOL) endpoints: 1) a 23-item physical distress level with scale score ranges from 23 to 92 [low score represents better QOL] 2)a 7-item psychological distress level with scale score ranges from 7 to 28[low score represents better QOL] 3)8-item activity level with scale score ranges from 8 to 32 [high score represents better QOL]; 1-item overall valuation of life with score range from 1 to 7 [low score represents better QOL].
Time Frame: Baseline until crossover treatment began (up to 82 months)
Population: Participants with RSCL at baseline and end of initial treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Gemcitabine Plus Docetaxel: gemcitabine 1000 mg/m2, intravenous, on Days 1 and 8 every 21 days plus docetaxel 75 mg/m2, intravenous, on Day 1 every 21 days. This treatment continues until progression of disease at which time crossover treatment begins.
- Docetaxel Plus Capecitabine: docetaxel 75 mg/m2, intravenous on Day 1 every 21 days plus capecitabine 1000 mg/m2, by mouth, twice a day, days 1-14, every 21 days. This treatment continues until progression of disease at which time crossover treatment begins.
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Number analyzed (Participants) | 117 | 118
units on a scale
  Baseline | 68.09 (25.103) | 72.32 (23.693)
  Change from Baseline | 2.42 (27.093) | -2.68 (26.685)
Statistical Analysis 1: Comparison: Gemcitabine Plus Docetaxel vs Docetaxel Plus Capecitabine; Test type: Superiority or Other; p = 0.801, Mixed Models Analysis

13. Secondary Outcome: Summary of Changes in Rotterdam Symptom Checklist by Treatment (Crossover Treatment)
Description: as for outcome 12
Time Frame: First day of crossover treatment until end of crossover treatment at trial discontinuation (up to 82 months)
Population: Participants with RSCL at baseline (conclusion of initial treatment)and end of crossover treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Capecitabine: capecitabine 1000 mg/m2, by mouth twice day, days 1-14 every 21 days until progression of disease at which time all treatment is discontinued.
Arm/Group | Capecitabine | Gemcitabine
Number analyzed (Participants) | 30 | 24
units on a scale
  Baseline | 75.00 (20.876) | 76.39 (17.663)
  Change from Baseline | -2.78 (21.029) | -0.69 (27.133)
Statistical Analysis 1: Comparison: Capecitabine vs Gemcitabine; Test type: Superiority or Other; p = 0.190, Mixed Models Analysis

ADVERSE EVENTS:
Description: A participant was randomized to comparator arm but treated with experimental treatment and thus included in the comparator arm ITT population (disposition and efficacy tables) and included in the experimental arm of treated population (AE tables). This results in an inconsistency between number of participants analysed and participant flow module.
Groups:
- Gemcitabine Plus Docetaxel: Initial treatment: Gemcitabine 1000 milligrams per meter squared (mg/m2), intravenous (IV) on Days 1 and 8 every 21 days plus docetaxel 75 mg/m2 IV on Day 1 every 21 days. This treatment continues until progression of disease (PD), at which time crossover treatment begins.
  Crossover treatment: capecitabine 1000 mg/m2 by mouth (PO) twice a day (BID), Days 1-14, every 21 days until PD at which time all treatment is discontinued.
Arm/Group | Gemcitabine Plus Docetaxel | Docetaxel Plus Capecitabine
Serious Adverse Events (participants affected / at risk) | 72/237 | 55/226
Other Adverse Events (participants affected / at risk) | 233/237 | 221/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Plus Docetaxel (N=237) | Docetaxel Plus Capecitabine (N=226)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (10) | 9 (9)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 6 (9) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 25 (38) | 7 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 4 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diverticulitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ruptured diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus of bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2)
Lethargy (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 5 (5)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Bilateral hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Phlebothrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Plus Docetaxel (N=237) | Docetaxel Plus Capecitabine (N=226)
Anaemia (Blood and lymphatic system disorders) | 113 (278) | 59 (110)
Leukopenia (Blood and lymphatic system disorders) | 86 (294) | 25 (53)
Neutropenia (Blood and lymphatic system disorders) | 193 (883) | 73 (216)
Thrombocytopenia (Blood and lymphatic system disorders) | 70 (152) | 6 (13)
Lacrimation increased (Eye disorders) | 15 (23) | 29 (38)
Abdominal pain (Gastrointestinal disorders) | 33 (42) | 30 (43)
Constipation (Gastrointestinal disorders) | 65 (100) | 49 (71)
Diarrhoea (Gastrointestinal disorders) | 111 (217) | 108 (221)
Dyspepsia (Gastrointestinal disorders) | 21 (28) | 28 (44)
Nausea (Gastrointestinal disorders) | 113 (233) | 118 (248)
Stomatitis (Gastrointestinal disorders) | 47 (92) | 60 (113)
Vomiting (Gastrointestinal disorders) | 71 (120) | 74 (134)
Asthenia (General disorders) | 45 (104) | 32 (61)
Chest pain (General disorders) | 15 (23) | 12 (13)
Fatigue (General disorders) | 129 (285) | 120 (224)
Mucosal inflammation (General disorders) | 38 (81) | 65 (117)
Oedema (General disorders) | 31 (77) | 27 (46)
Oedema peripheral (General disorders) | 54 (90) | 44 (67)
Pain (General disorders) | 25 (45) | 18 (31)
Pyrexia (General disorders) | 60 (93) | 33 (38)
Rigors (General disorders) | 15 (22) | 9 (9)
Candidiasis (Infections and infestations) | 5 (9) | 12 (14)
Upper respiratory tract infection (Infections and infestations) | 17 (21) | 8 (8)
Urinary tract infection (Infections and infestations) | 13 (19) | 11 (11)
Alanine aminotransferase increased (Investigations) | 28 (42) | 13 (19)
Aspartate aminotransferase increased (Investigations) | 21 (31) | 14 (22)
Weight decreased (Investigations) | 16 (23) | 10 (14)
Anorexia (Metabolism and nutrition disorders) | 59 (122) | 59 (92)
Dehydration (Metabolism and nutrition disorders) | 21 (24) | 22 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (47) | 15 (21)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (22) | 12 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (16) | 14 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 (60) | 39 (62)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (34) | 23 (31)
Bone pain (Musculoskeletal and connective tissue disorders) | 21 (29) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 46 (105) | 33 (62)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (42) | 25 (31)
Dizziness (Nervous system disorders) | 21 (24) | 19 (32)
Dysgeusia (Nervous system disorders) | 32 (50) | 29 (39)
Headache (Nervous system disorders) | 41 (53) | 32 (38)
Peripheral sensory neuropathy (Nervous system disorders) | 78 (133) | 83 (141)
Depression (Psychiatric disorders) | 16 (21) | 9 (10)
Insomnia (Psychiatric disorders) | 31 (38) | 30 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 54 (92) | 45 (55)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 (81) | 37 (51)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 (26) | 11 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 86 (120) | 98 (127)
Erythema (Skin and subcutaneous tissue disorders) | 10 (10) | 15 (19)
Nail disorder (Skin and subcutaneous tissue disorders) | 38 (70) | 67 (118)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (20) | 129 (370)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (16) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 59 (82) | 32 (44)
Hypotension (Vascular disorders) | 12 (13) | 6 (6)
Lymphoedema (Vascular disorders) | 14 (24) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days